CLINICAL TRIAL: NCT06549803
Title: A Study on Comparison of Postoperative Outcome Between Conventional Skin Stapling and Tissue Adhesive (2-octyl Cyanoacrylate) for Skin Closure in Colorectal Cancer
Brief Title: Comparison of Method for Skin Closure in Colorectal Cancer.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yoon Suk Lee (Other)
Collaborators: Dalim BioTech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yoon Suk Lee, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC21EISI0608
Record Dates: First submitted 2024-07-03; First posted 2024-08-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-08

CONDITIONS: Surgical Site Infection; Colorectal Cancer
Keywords: colorectal cancer; skin adhesive bond; skin stapling
MeSH Terms: conditions — Surgical Wound Infection; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Skin adhesive bond (Experimental): a group which skin closure was performed using Leukosan Adhesive skin bond
  Interventions: Device: skin bond
- skin stapler (Active Comparator): a group which skin closure was performed using skin stapler
  Interventions: Device: skin stapler

INTERVENTIONS:
Device: skin bond — In the skin bond group, fascia closure is performed for incision sites of 10 mm or more, and skin bond is sufficiently applied after subcuticular suture.
  For incision sites less than 10 mm, subcuticular closure is performed without closing the fascia, and then skin bond is applied.
  Arms: Skin adhesive bond
Device: skin stapler — In the skin stapler group, fascia closure is performed on incision sites larger than 10 mm, and the skin is closed at 2-3 mm intervals using a stapler.
  For incision sites less than 10 mm, skin closure is performed using a skin stapler without closing the fascia.
  Arms: skin stapler

SUMMARY:
Compared to tissue adhesives and skin stapling devices, tissue adhesives are reported to have advantages in terms of wound infection and cost competitiveness. However, there have been no prospective randomized studies focusing on wound infection rates and cost competitiveness between skin stapling devices and tissue adhesives in colorectal cancer surgery.

In colon cancer surgery, it is still unclear which skin suturing method has advantages such as lower postoperative wound infection rate and price competitiveness. The purpose of this study is to compare clinical outcomes, including wound infection rates and cost-effectiveness, between two different wound closure methods for colorectal cancer.

DETAILED DESCRIPTION:
The primary purpose of the study is to compare and analyze the incidence of surgical site infection within 30 days after surgery in each group when tissue adhesive was applied and when skin stapling device was applied.

The purpose of the secondary study is to compare the clinical results after surgery by analyzing cost-effectiveness, pain level, and satisfaction after surgery between existing skin stapling and tissue adhesive for colon cancer patients.

Post-operative wound infection rate, cost (material costs of staplers, adhesives, material costs and service fees for disinfecting wounds occurring in the week after surgery), sex, age, BMI (body mass index), ASA (Anesthesiologists category), past history (diabetes, smoking history) , past abdominal surgery history), cancer stage, pre- and post-operative blood test results (WBC, CRP), biopsy results (cancer type), surgery time, pain on the 1st and 3rd days after surgery (VAS), length of stay, postoperative complications , compare the postoperative results of satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* underwent elective colorectal surgery
* aged 19 to 80 years
* ASA (American Society of Anesthesiologists) score: 1, 2
* surgical approach such as laparoscopic or Robotic Xi platform

Exclusion Criteria:

* ASA score above 3
* Aged over 80 years
* underwent combined surgery for other organ resection
* uncontrolled DM

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of surgical site infection within 30 days after surgery | through study completion, an average of 1 year
  Comparative analysis of the frequency of surgical site infection up to 1 month after surgery in each group when tissue adhesive was applied and when skin stapling device was applied.

SECONDARY OUTCOMES:
Postoperative pain score | through study completion, an average of 1 year
  Post-operative pain score by VAS score were measured and compared with each other by understanding various factors through cost-effectiveness analysis, pain level, satisfaction, etc. after surgery between existing skin stapling and tissue adhesive for colon cancer patients.
Postoperative wound dressing cost | through study completion, an average of 1 year
  Postoperative wound dressing cost between existing skin stapling and tissue adhesive for colon cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Suk Lee, M.D.,Ph.D, Study Chair — Department of Surgery, Seoul St.Mary's hospital
Locations (1):
- Seoul St.Mary's hospital, the Catholic university of Korea, Seoul, Seocho, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yahara S, Kishimoto Y. Characterization of alkylgalactolipids from calf brain by high performance liquid chromatography. J Neurochem. 1981 Jan;36(1):190-4. doi: 10.1111/j.1471-4159.1981.tb02394.x. PMID 7463045